CLINICAL TRIAL: NCT02360241
Title: LPRobacus: Light Needle Positioning Robot Under MRI Guidance
Brief Title: Light Needle Positioning Robot Under MRI Guidance
Acronym: LPRobacus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: TIMC-IMAG (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: DCIC 14-36
Record Dates: First submitted 2015-01-12; First posted 2015-02-10 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-10

CONDITIONS: Magnetic Resonance Imaging; Robotic Surgical Procedures
MeSH Terms: interventions — Robotic Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Robot (Experimental): A robot will be used and it's position will be evaluated
  Interventions: Device: Robot

INTERVENTIONS:
Device: Robot — Use of the robot to locate the fictional needle

SUMMARY:
This study aim is to evaluate the needle positioning precision, compared to the real path planned by the physician on healthy voluntaries, by positioning a fictional needle, without inserting it.

Additionally, this study will evaluate:

* the robot precision,
* the robot detection robustness,
* the software and device ergonomics,
* the device security.

ELIGIBILITY:
Inclusion Criteria:

* person over 18 years old,
* person with height is under 1m90,
* person with abdomen height is under 28 cm,
* person with abdomen width is between 26 cm to 50 cm,
* person able to hold his breath during 30 seconds,
* person affiliated to social security or similarly regime,
* signed consent for participation in the study.

Exclusion Criteria:

* person with a contraindication for abdomen MRI,
* claustrophobic person,
* protected person referred to in Articles L1121-5 to L1121-8 of the Code of Public Health

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Amount of needle positioning needed to reach the real path wanted, with a 5mm precision (cylinder diameter including the path defined by the two skin marker and the need axe). | 1hour20minutes
  evaluate the real needle positioning precision: the robot effectiveness

SECONDARY OUTCOMES:
Number of time in percentage of failed robot use. | 1hour20minutes
  evaluate the robot detection robustness
Number of time in percentage of failed fixation of the robot over the patient. | 1hour20minutes
  match of the robot fixation system
Score from a qualitative evaluation scale of the healthy voluntary discomfort during robot use and the score from a scale of the physician satisfaction (girth, ease, speed). | 1hour20minutes
  device and software ergonomics
Number of time in percentage that the robot was stopped (voluntary/dysfonctionnement) during its use | 1hour20minutes
  Device security

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Bricault, PhD, Pr, Principal Investigator — echipon@chu-grenoble.fr
Locations (1):
- University Hospital Grenoble, Grenoble, Isère, France

REFERENCES:
- See also: Website of the Grenoble clinical investigation center - Technological Innovation — http://www.cic-it-grenoble.fr/
- See also: Website of TIMC-IMAG laboratory — http://www-timc.imag.fr/